CLINICAL TRIAL: NCT02427607
Title: An Open-label Extension Study to Evaluate the Safety and Tolerability of Perampanel (E2007) Administered as an Adjunctive Therapy in Epilepsy Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-J000-341
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Results first posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-09

CONDITIONS: Epilepsy
Keywords: Epilepsy; Perampanel
MeSH Terms: conditions — Epilepsy | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perampanel (Experimental): Participants started the study with the dose that they were receiving at the end of their participation in the previously participated Study E2007-G000-332 (Study 332) [NCT02307578]. Doses of perampanel were allowed to be adjusted based on clinical judgment. A minimum perampanel dose of 2 milligram (mg) per day was required to continue in the study. The maximum daily dose of perampanel permitted was 12 mg per day.
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — Perampanel 2 mg tablets. Doses of perampanel can be adjusted based on clinical judgment. A minimum perampanel dose of 2 mg per day is required to continue in the study. The maximum daily dose of perampanel permitted will be 12 mg per day.
  Other Names: Fycompa; E2007

SUMMARY:
To evaluate the safety and tolerability of perampanel given as an adjunctive therapy in participants with epilepsy. This study will be continued until perampanel is commercially available.

ELIGIBILITY:
Inclusion Criteria

1. Participants participating in the designated perampanel study as below, and who in the opinion of the investigator continue to benefit from treatment with perampanel Designated perampanel study: E2007-G000-332 (NCT01393743) (with at least 52 weeks of total exposure to perampanel).
2. Provide written informed consent/assent signed by participant or legal guardian prior to entering the study or undergoing any study procedures. If the written informed consent is provided by the legal guardian because the participant is unable to do so, a written or verbal assent from the participant must also be obtained.
3. Female participants of childbearing potential must agree for the duration of the study and for a period of at least 1 month following the last dose of perampanel to be abstinent or to commit to the consistent and correct use of a medically acceptable method of birth control (eg, a double-barrier method [condom plus spermicide, condom plus diaphragm with spermicide]).

Exclusion Criteria

1. Participants residing in countries where perampanel is commercially available with respect to the indication or formulation of the designated perampanel study.
2. Female participants who are nursing, pregnant, or planning to become pregnant.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2016-09-21 (Actual); Study Completion 2016-11-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Japan (8):
  - Matsuyama, Ehime
  - Sapporo, Hokkaido
  - Inashiki-gun, Ibaraki
  - Uji, Kyoto
  - Sakai, Osaka
  - Matsue, Shimane
  - Nerima-Ku, Tokyo
  - Niigata

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 8 centers in Japan during the period of 12 May 2015 to 21 Sep 2016. E2007-J000-341 is an open-label extension of E2007-G000-332.
Period: Overall Study
Arm/Group | Perampanel
Started | 7
Completed | 6
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who signed informed consent and received at least one dose of study drug, and had at least one post-dose safety assessment in Study 341.
Arm/Group | Perampanel
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.3 (19.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) as a Measure of Safety and Tolerability of Perampanel
Description: Safety was assessed by monitoring adverse events (AEs), withdrawal from treatment, clinical laboratory tests (chemistry), vital signs, and weight. TEAEs were defined as AEs that emerged from the first dose of study drug to the last visit of Study 341 or on or after 30 days since the last dose of study drug in Study 341, whichever comes later, having been absent at pretreatment (Baseline of Study 332). A markedly abnormal clinical chemistry laboratory value was defined as a laboratory result that worsened in severity to meet modified National Cancer Institute (NCI) toxicity criteria of Grade 2 or higher on treatment. Treatment-related TEAEs were defined as AEs that were considered by the investigator to be possibly or probably related to study treatment. SAEs were defined as any untoward medical occurrence that at any dose; resulted in death, disability/incapacity, birth defect, required inpatient hospitalization or prolongation of existing hospitalization, or was life-threatening.
Time Frame: From first dose of study drug until perampanel was commercially available, up to approximately 1 year 5 months
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Perampanel
Number analyzed (Participants) | 7
Participants
  Non-Serious TEAEs | 6
  Treatment-related TEAEs | 0
  Severe TEAEs | 0
  TEAEs leading to study drug dose adjustment | 0
  Serious TEAE | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug until perampanel was commercially available, up to approximately 1 year 5 months
Description: Treatment-emergent adverse events (TEAEs) and serious adverse events were reported. The safety analysis set included all participants who signed informed consent and received at least one dose of study drug, and had at least one post-dose safety assessment in Study 341. TEAEs were AEs that emerged from first dose of study drug to last visit of Study 341 or on or after 30 days since the last dose of study drug in Study 341, whichever came later, having been absent at Baseline of the Study 332.
Arm/Group | Perampanel
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 6/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (N=7)
Nasopharyngitis (Infections and infestations) | 3
Influenza (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other